CLINICAL TRIAL: NCT06203925
Title: Hepatitis C Virus Self-testing (HCVST) in Sexual and Gender Minorities in Rio de Janeiro (Brazil): Distribution and Uptake of HCV Testing Using Internet Technology and Evaluation of Usability of HCVST
Brief Title: Hepatitis C Virus Self-testing (HCVST) in Sexual and Gender Minorities in Rio de Janeiro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: World Health Organization (Other); UNITAID (Other)
Responsible Party: Sponsor
Other Study IDs: 69747223.4.0000.5262
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus self-test; Sexual and Gender Minorities
MeSH Terms: conditions — Hepatitis C; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Primary Study: The study will be a cohort study. Adult SGM living in the metropolitan area of Rio de Janeiro who voluntary want to perform HCV testing ordered through a web-based platform will be eligible for this study. SGM will be defined by gay, bisexual and other cisgender MSM, TGW, transgender men, and gender nonbinary/diverse individuals.
  Interventions: Diagnostic Test: Hepatitis C virus self-test (oral fluid HCVST); Diagnostic Test: Hepatitis C virus self-test (blood-based HCVST)
- Ancillary Study: The study will be a cross-sectional study. Adult MSM or TGW attending a presential visit for PrEP (initiation or follow-up) at INI/FIOCRUZ will be eligible for this study.
  Interventions: Diagnostic Test: Hepatitis C virus self-test (oral fluid HCVST); Diagnostic Test: Hepatitis C virus self-test (blood-based HCVST)

INTERVENTIONS:
Diagnostic Test: Hepatitis C virus self-test (oral fluid HCVST) — The participant will be able to choose between oral-fluid or blood-based HCVST. The package will include an HCV OraQuick ® HCV Self-Test kit, (OraSure Technologies, Inc, Bethlehem, PA) or a Wondfo® HCV Self-Test (Guangzhou, P.R. China) at Primary Study.
  At Ancyllary study, the individuals attending PrEP consultations at INI/FIOCRUZ will be invited to perform HCVST using blood-based and oral-fluid kits.
  Other Names: OraSure Technologies, Inc, Bethlehem, PA
Diagnostic Test: Hepatitis C virus self-test (blood-based HCVST) — The participant will be able to choose between oral-fluid or blood-based HCVST. The package will include an HCV OraQuick ® HCV Self-Test kit, (OraSure Technologies, Inc, Bethlehem, PA) or a Wondfo® HCV Self-Test (Guangzhou, P.R. China) at Primary Study. At Ancylary Study, the individuals attending PrEP consultations at INI/FIOCRUZ will be invited to perform HCVST using blood-based and oral-fluid kits.
  Other Names: Wondfo® HCV Self-Test (Guangzhou, P.R. China)

SUMMARY:
Sexual and gender minorities (SGM), such as gay, bisexual and other men who have sex with men (MSM) and transgender women (TGW), are at high risk of HCV infection. A recently released guideline by the WHO recommended HCVST to scale-up HCV screening. However, data on delivery-services of HCVST kits and uptake of HCV testing using HCVST remain scarce in Latin American countries. Additionally, data on the usability of HCVST in MSM/TGW, especially blood-based tests, still lacking in Brazil. To evaluate the uptake of HCV testing by the strategy of using HCVST ordered by the internet and delivery by the post in key populations (SGM) living in the metropolitan region of Rio de Janeiro (Brazil). Additionally, an Ancillary study will assess the usability of different kits of HCVST in MSM/TGW using PrEP.

Study Design and Population: This protocol will be composed of two studies that will be conducted in parallel. The primary study will be a cohort study in which SGM ≥ 18 years old living in the metropolitan area of Rio de Janeiro who request HCVST will be included. The Ancillary study will be a cross-sectional study where adult MSM or TGW attending a presential visit for PrEP (initiation or follow-up) at INI/FIOCRUZ will be eligible for this study. The investigators estimate that 3,000 persons will request home-delivery of HCVST (Primary study) and 250 participants will be included in the Ancillary study.Study Design and Population: This protocol will be composed of two studies that will be conducted in parallel. The primary study will be a cohort study in which SGM ≥ 18 years old living in the metropolitan area of Rio de Janeiro who request HCVST will be included. The Ancillary study will be a cross-sectional study where adult MSM or TGW attending a presential visit for PrEP (initiation or follow-up) at INI/FIOCRUZ will be eligible for this study. The investigators estimate that 3,000 persons will request home-delivery of HCVST (Primary study) and 250 participants will be included in the Ancillary study.

Methods: For the Primary Study, a web-based platform will be built for this project and an educational campaign will be developed in dating apps to encourage HCV testing. The web platform will contain modules with information on HCV infection and a log-in to request HCV self-tests that can be delivered by the post or collected in the centralized pharmacy for HCV testing. People will be encouraged to report their HCVST results in the online platform. People with positive HCV antibody will be linked-to-care for HCV infection confirmation and treatment initiation. For the Ancillary Study, MSM/TGW attending presential visits for PrEP at INI/FIOCRUZ will be invited to perform HCVST (blood-based and oral fluid tests) under supervision of a trained healthcare worker. Participants will read written instructions and watch a video explaining the procedures step-by-step for HCVST. A second HCV test using the same kit will be performed by the healthcare worker for concordance analysis. People with positive HCV antibodies will be linked to HCV infection confirmation and treatment initiation.

Data analysis: Descriptive statistical analysis will be used to evaluate the characteristics of people seeking HCVST, participant's preferences, uptake of HCV testing using self-test kits and internet technologies, as well as acceptability, usability and result interpretation of HCVST in a sub-sample of participants. Ethical considerations: Locally, ethics approval will be obtained from the INI/FIOCRUZ. International ethics clearance will be obtained from the World Health Organization Ethics Review Committee (WHO ERC). All participants will be informed of risks and benefits of the procedures and that their participation is voluntary. All participants will be required to sign the informed consent (an online agreement for Primary Study) as required by Brazilian regulations to participate in research studies. All data collected will respect The Brazilian General Data Protection Law (Law nº 13.709/2018).

DETAILED DESCRIPTION:
Chronic hepatitis C is a major health issue in Brazil where it is estimated that up to 650,000 people are living with HCV infection. Despite the availability of rapid tests as well as universal access to safe and highly effective drugs for HCV treatment for free of charge, the HCV HCV continuum of care remains unsatisfactory. HCV transmission due to sexual activities are increasing in Brazil, especially among young men. It is well known that MSM and/or TGW are at high risk for HCV infection. HCV infection in these key populations might occur mainly in the context of traumatic sex practices that increase the risk of blood-blood contact. The use of drug prior to or during sex (chem-sex) might be associated with HCV infection. Few studies have reported the prevalence of HCV infection among SGM in Brazil. Firstly, a single center study that included a limited sample (n=522) using Respondent-Driven Sampling reported a prevalence of anti-HCV positive of 1.3% (95%CI: 0.3-5.5) in MSM in Central region. All people with anti-HCV positive reported high-risk sexual behaviors, condomless use at anal intercourse and frequent chem-sex [39]. More recently, the prospective, single-arm, open-label, multicentre PrEP implementation study conducted in Brazil (14 sites), Mexico (4 sites), and Peru (10 sites) included 9,509 HIV-negative MSM and TGW for daily oral initiation of PrEP. Prevalence of hepatitis C increased from the enrolment to week-52 among participants from Mexico and Peru, cisgender men, and those aged 25-30 years. In Brazil (n=3,928), the prevalence of HCV infection was 0.34% (95%CI 0.16-0.52) and 0.58% (95%CI 0.24-0.91) at enrolment and week-52, respectively [40]. Similarly, a Brazilian study reported an HCV prevalence of 0.66% (anti-HCV positive in 340 from 51,486 tests) in key populations (MSM, transgender people, people who inject drugs, and sex workers) in Curitiba (Southern region) [24] Similar to other countries, HIV coinfection and injection drug use have been associated with increased risk of HCV infection/reinfection in Brazil. Prevalence of HCV infection (2.7%) was mostly associated with injection drug use in the last year [OR=10.33 (95%CI 4.74-22.52)] and HIV infection [OR=4.74 (95%CI 1.82-12.36)] in Brazilian men prisoners (n=2,848)[41].

Large scale screening for hepatitis C in high-risk people and linkage-to-care are cornerstones towards to HCV elimination. HCVST can decrease the barriers to traditional testing by increasing convenience and privacy. Lesson learned with HIVST can be informative and suggest that this new/additional testing approach may help to increase HCV testing and linkage to care and treatment. A recently released guideline by the WHO recommended HCVST to scale-up HCV screening [6]. In brief, this guideline recommends that HCVST should be offered as an additional approach to facility-based HCV testing. Additionally, HCVST needs to be followed by confirmation of viremic infection (HCV-RNA), and linkage-to-treatment, and HCVST service delivery should be adapted to local context, which includes community preferences. However, the usability of HCVST kits, cost-effective, non-discriminatory and inclusive service delivery and optimal position of HCVST in national HCV programs must be addressed. Stigma is an important element in the experience of living with chronic HCV infection, especially in SGM persons. This stigma impacts in healthcare access and uptake as well as health outcomes. The use of HCVST can help to mitigate the stigma along the HCV continuum of care. Additionally, the immediate linkage to care after a positive HCVST using telehealth might reduce mental distress from positive results.

Recent studies have evaluated the usability, acceptability, and rates of interpretation of results from different kits (blood-based and oral fluid) of HCVST worldwide. Few studies reported high acceptability and usability of oral-fluid HCVST in key populations (mostly MSM), especially in the USA, European countries and Asia. However, data on delivery-services of HCVST kits and uptake of HCV testing using HCVST remain scarce in Latin American countries. Additionally, data on the usability of HCVST in MSM/TGW, especially blood-based tests, still lacking in Brazil. This study will evaluate the uptake of HCV testing by the strategy of using HCVST that would be able to be ordered by the internet and delivery by the post in key populations (SGM) living in the metropolitan region of Rio de Janeiro (Brazil). Additionally, a sub-study will assess the acceptability, usability and result interpretation of different kits of HCVST in MSM/TGW using PrEP in a reference center in Rio de Janeiro (Brazil).

This project will assess operational research priorities about HCVST in Brazil. The investigators expect to fulfill gaps of knowledge on product optimization (acceptability and usability of blood-based and oral fluid HCVST kits), service delivery and linkage pathways to confirmatory testing and treatment after reactive HCVST results in one of the largest agglomerations worldwide, such as the metropolitan area of Rio de Janeiro (Brazil). The investigators expect to increase HCV testing by using an online platform to inform about HCV infection where people will be able to order HCVST that can be delivered by the post. Additionally, our strategy will include an offer of HIVST with HCVST (combo HIV/HCVST) to increase interest for HCV testing and a massive advertising campaign in dating-apps used by SGM (e.g. Grindr, Scruff and Hornet). In addition, the investigators expect that HCVST will be highly accepted and easy to be performed among PrEP users in Rio de Janeiro (Brazil).

This protocol will be composed by a Primary Study and an Ancillary Study that will be conducted in parallel.

OBJECTIVES:

The Primary Study will assess HCVST using internet-technologies among SGM. The main hypothesis of the Primary Study is that HCVST ordered in an online platform and delivered by the post will increase HCV testing uptake among SGM.

The Ancillary Study will assess the acceptability and usability of different kits of HCVST in MSM/TGW under PrEP. The main hypothesis of the Ancillary Study is that blood-based and oral fluid HCVST will be well accepted and easily to be performed among MSM/TGW under PrEP in a referral center in Rio de Janeiro (Brazil)

2.1. Overall objectives Overall objective of the Primary Study: To evaluate the uptake of HCV testing using HCVST ordered through a web-based platform among SGM living in Rio de Janeiro (Brazil) Overall objective of the Ancillary Study: To evaluate the acceptability, usability, results interpretation and participant's perspectives of HCVST with blood-based and oral-fluid kits among MSM and TGW who are attending a PrEP visit in a reference center in Rio de Janeiro (Brazil).

2.2 Specific objectives

Specific objectives of the Primary Study:

1. To describe socio-demographic characteristics of people seeking HCV self-testing
2. To evaluate preference for oral fluid or blood-based HCV self-tests
3. To evaluate the proportion of people using home-based delivery vs pick up of HCV self-tests
4. To evaluate the proportion of people reporting HCV self-test results
5. To evaluate the proportion of people attending a consultation when HCV self-test is reactive or invalid
6. To evaluate the knowledge of SGM about HCV infection and/or treatment
7. To evaluate cost per case of HCV infection detected using HCV self-testing and internet technologies
8. To evaluate the proportion of people with reactive HCVST who had HCV-RNA test for confirmation and who started HCV treatment (linkage to HCV continuum of care)
9. To evaluate the proportion of people who ordered HCVST to receive an HIVST kit

Specific objectives of the Ancillary Study:

1. To describe socio-demographic characteristics of people under PrEP performing HCVST
2. To evaluate the proportion of people who correctly perform HCVST
3. To evaluate the proportion of people who do not need assistance to correctly perform HCVST
4. To evaluate the proportion of people who correctly report HCVST results (re-read by a trained healthcare worker)
5. To evaluate the concordance of HCVST with re-testing by a trained healthcare worker
6. To evaluate the preference for oral-fluid or blood-based HCVST kits
7. To evaluate the proportion of people attending a consultation when HCV self-test is reactive or invalid
8. To evaluate the knowledge of people under PrEP about HCV infection and/or treatment
9. To evaluate cost per case of HCV infection detected using HCVST in PrEP users
10. To evaluate the proportion of people with reactive HCVST who had HCV-RNA test for confirmation and who started HCV treatment (linkage to HCV continuum of care)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old with knowledge of the Portuguese language
2. Self-identification as gay, bisexual and other cisgender MSM, TGW, transgender men, and gender nonbinary/diverse individuals
3. Reported residence in the metropolitan area of Rio de Janeiro (municipalities of Rio de Janeiro, Duque de Caxias, São João de Meriti, Belford Roxo, Nilópolis, Mesquita, Nova Iguaçu, Queimados, Japeri, Paracambi, Seropédica, Itaguaí, Magé, Guapimirim, Niterói, São Gonçalo, Itaboraí, Seropédica, Rio Bonito, Tanguá and Maricá)

Exclusion Criteria:

1. Unable or not willing to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification as gay, bisexual and other cisgender MSM, TGW, transgender men, and gender nonbinary/diverse individuals
Study Population: Primary Study:
  Participants reported residence in the metropolitan area of Rio de Janeiro (municipalities of Rio de Janeiro, Duque de Caxias, São João de Meriti, Belford Roxo, Nilópolis, Mesquita, Nova Iguaçu, Queimados, Japeri, Paracambi, Seropédica, Itaguaí, Magé, Guapimirim, Niterói, São Gonçalo, Itaboraí, Seropédica, Rio Bonito, Tanguá and Maricá)
  Ancillary Study:
  2. Self-identification as MSM or TGW 3. Presential visit for PrEP (initiation or follow-up) at INI/FIOCRUZ
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of SGM living in Rio de Janeiro (Brazil) who requested an HCVST kit through a web-based platform | 1 month
  Captured datas obtained from a web-based plataform
Number of SGM living in Rio de Janeiro (Brazil) who received and performed the test. | 1 month
  Captured datas obtained from a web-based plataform
Proportion of MSM/TGW who correctly performed HCVST with oral-fluid and blood-based kits without assistance of a healthcare worker | 1 day
  Captured datas obtained from a web-based plataform

SECONDARY OUTCOMES:
Socio-demographic characteristics through the data obtained from the study. | 2 months
  - Socio-demographic characteristics of SGM seeking HCVST in Rio de Janeiro
Type-preference test through the data obtained from the study. | 2 months
  - Proportion of type-preference [oral fluid vs blood-based; home-based delivery vs pick-up] for HCVST
Participants who reported Easy test. | 2 months
  - Proportion of people who reported HCVST as "Easy/Very Easy" to be performed
Possible outcomes through the data obtained from the study. | 2 months
  - Proportion of people reporting HCVST results at the web-based platform
Participants through the data obtained from the study. | 2 months
  - Proportion of people correctly interpreting HCVST results
Participants who attending a consultation through the data obtained from the study. | 2 months
  - Proportion of people attending a consultation after an HCVST result as reactive or invalid
Prevalence of reactive HCV through the data obtained from the study. | 2 months
  - Prevalence of reactive HCV antibody by HCVST in SGM in Rio de Janeiro
Cost per identification through the data obtained from the study. | 2 months
  - Cost per identification of chronic hepatitis C individual using HCVST
Particiopants who used telehealth through the data obtained from the study. | 2 months
  - Proportion of people who accepted and used telehealth for linkage-to-care for HCV infection
Socio-demographic characteristics of MSM/TGW through the data obtained from the study. | 1 month
  - Socio-demographic characteristics of MSM/TGW who agreed to perform HCVST
Participants who report the test through the data obtained from the study. | 1 month
  - Proportion of people who correctly report HCVST results (using re-reading by a trained healthcare worker as the reference)
Participants who needed help from a healthcare. | 1 month
  - Proportion of case where results of HCV re-testing by a trained healthcare worker was concordance with HCVST using the same kit
Preference for tests | 1 month
  - Proportion of type-preference [oral fluid vs blood-based] for HCVST
Easy test | 1 month
  - Proportion of people who reported HCVST as "Easy/Very Easy" to be performed
Participants who needed a consultation. | 1 month
  - Proportion of people attending a consultation after an HCVST result as reactive or invalid
Positive participants | 1 month
  - Prevalence of reactive HCV antibody by HCVST in MSM/TGW attending a PrEP visit
Cost for using the test | 1 month
  - Cost per identification of chronic hepatitis C individual using HCVST in a PrEP scenario
Positive participants with HCV-RNA | 1 month
  - Proportion of people with reactive HCVST who had HCV-RNA test for confirmation and who started HCV treatment (linkage to HCV continuum of care)

CONTACTS AND LOCATIONS:
Locations (1):
- Evandro Chagas National Institute of Infectious Diseases, Rio de Janeiro, Rio de Janeiro/RJ, Brazil

IPD SHARING:
Plan to Share IPD: No
There is a risk of loss of participant confidentiality and there is no authorization from the ethics committee to make individual data available. All data will be made available through scientific publications.